CLINICAL TRIAL: NCT02816723
Title: Improving Brain Health in Older Veterans: A Mindfulness Training Pilot Study
Brief Title: Mindfulness Training in Healthy Older Veterans
Acronym: MTGHOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2398-P
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Aging
Keywords: mindfulness; aging; Veterans
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness (Experimental): mindfulness/meditation/movement training
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Brain Health (Active Comparator): Brain Health education class
  Interventions: Behavioral: Brain Health

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — mindfulness/meditation/movement training
  Other Names: MBSR
  Arms: Mindfulness
Behavioral: Brain Health — Brain Health Education
  Arms: Brain Health

SUMMARY:
Evidence shows the positive effects of Brain Health & Wellness classes in younger individuals. The proposed study investigates the usefulness of these classes in older Veterans aged 50-85. We hope to show that such classes can lead to improvements in both thinking skills as well as stress levels.

DETAILED DESCRIPTION:
The expansion of the aging Veteran population, in addition to the frequent presence of comorbidities (e.g., PTSD and TBI) that exacerbate age-associated cognitive and health declines, has generated substantial interest in interventions that promote brain health in older Veterans. A growing body of evidence shows the positive effects of Brain Health & Wellness classes on brain health in younger and middle-aged adults, thus training might be able to enhance brain health in older Veterans and offset age-related declines. Such training holds particular promise in enhancing areas of cognition that are especially susceptible to aging processes (e.g. attention and executive control), potentially through multiple mechanistic pathways. It is in many respects a cognitive exercise and may strengthen neural networks involved in such processes. Additionally, there is evidence for further facilitating brain health in other ways related to, for instance, altering the stress response. Currently, there is little information regarding the potential brain health benefits in older adults. As a first step to understanding these potential beneficial effects in Veterans, the aim of the proposed pilot study is to evaluate the acceptability, feasibility and potential efficacy of two Brain Health & Wellness classes in healthy older Veterans through a randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be Veterans age 50-85

Exclusion Criteria:

* moderate or severe TBI
* active alcohol or drug dependence or abuse by DSM-5 criteria (within previous 30 days)
* positive urine drug screen for illicit substances
* history of schizophrenia
* ADHD
* learning disability
* dementia
* Mild Cognitive Impairment and/or other psychiatric disturbances not including PTSD and/or depression
* participants with a history of psychiatric hospitalization (last five years)
* suicide attempt (last five years)
* imminent risk for suicidal or homicidal behavior, or severe medical illness requiring treatment will be excluded
* subjects with a history of neurological diagnosis, e.g.,:

  * brain tumor
  * clinical stroke
  * seizure
* Mini-Mental Status Exam score below 19 (suggesting moderate/severe cognitive impairment, a contraindication to MBSR participation) will be excluded

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana V. Baldo, PhD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness | Brain Health
Started | 30 | 30
Completed | 24 | 28
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness: Mindfulness-based Stress Reduction (MBSR): The MBSR group meets once per week for 2½ hours, with a day-long retreat in the 6th week of the 8-week program. Participants are instructed in mindfulness practice in the form of sitting meditation, body awareness, yoga, mindful movement, and informal mindfulness practices of daily life (e.g., eating, communicating, working, coping). The day-long retreat includes a review of class material, more lengthy meditation and yoga practice, as well as a group lunch. Between classes, patients enhance their participation by practicing at home with meditation CDs, homework assignments, and readings from the course materials and manual. Home practice is tracked with pre-made log sheets on which participants record the number of hours engaged in practice at home.
- Brain Health: Brain Health education class:
  The Brain Health class is matched for the same number of hours, instructor, schedule (including day-long retreat), homework, and home practice as that of the MBSR class. The class provides background and education about brain-behavior relationships and discusses how brain injuries can disrupt various aspects of cognition, such as memory and attention. There are also units on nutrition and sleep, including strategies for successful aging. To control for the yoga/movement portion of the MBSR class, the Brain Health class also includes simple chair exercises, such as stretching and reaching. The day-long retreat includes review of class topics, video documentaries on these topics, and a group lunch. The Brain Health class matches MBSR intervention for critical process elements such as clinician interaction, social interaction with the group, movement, schedule, and homework activities, without the inclusion of a meditative/mindfulness component.
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Brain Health | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 20 | 26 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (7.6) | 74.1 (7.3) | 73.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 17 | 22 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52
Number of years of formal education, 0-20 years [Mean (Standard Deviation); unit: years] — The number of years of formal education was a self-report measure. Participants told examiner what level of schooling they had completed, e.g. 12 years = high school completion and 16 years = college completion.
  years | 16.2 (2.2) | 16.9 (2.6) | 16.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Geriatric Depression Scale Change Score
Description: Participants' scores on the Geriatric Depression Scale were collected within 2 weeks before the intervention and again within 2 weeks after the intervention. This outcome measure represents the change in score in Geriatric Depression Scale: pre-intervention score minus post-intervention score. The maximum Geriatric Depression Scale score is 30, and the minimum score is 0. Higher scores on the Geriatric Depression Scale indicate more depressive symptoms, so worse outcome. However, since we are analyzing a change in the Geriatric Depression Scale score of pre- minus post-intervention, a larger change score for a particular arm indicates a greater degree of improvement.
Time Frame: Baseline (within two weeks pre-intervention) and Outcome at 2 months (within 2 weeks post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness | Brain Health
Number analyzed (Participants) | 24 | 28
score on a scale | .89 (1.79) | 0.50 (.21)

2. Primary Outcome: State-Trait Anxiety Inventory (STAI) Change Score
Description: Participants' scores on the State-Trait Anxiety Inventory (STAI) were collected within 2 weeks before the intervention and again within 2 weeks after the intervention. This outcome measure represents the change in score in State-Trait Anxiety Inventory: pre-intervention score minus post-intervention score. The maximum STAI score is 80, and the minimum score is 20. Higher scores on the STAI indicate more anxiety symptoms, so worse outcome. However, since we are analyzing a change in the STAI score of pre- minus post-intervention, a larger change score for a particular arm indicates a greater degree of improvement.
Time Frame: Baseline (within two weeks pre-intervention) and Outcome at 2 months (within 2 weeks post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness | Brain Health
Number analyzed (Participants) | 24 | 28
units on a scale | .06 (.22) | 2.75 (1.21)

3. Secondary Outcome: Repeatable Battery for Neuropsychological Status (RBANS) Total Scaled Change Score
Description: Participants' scores on the Repeatable Battery for Neuropsychological Status (RBANS) were collected within 2 weeks before the intervention and again within 2 weeks after the intervention. The maximum total scaled score is 160, and the minimum score is 40, where higher scores are better. This outcome measure represents the change in total scaled score on the RBANS: post-intervention score minus pre-intervention score. A higher change score for a particular arm indicates a greater degree of improvement.
Time Frame: Baseline (within two weeks pre-intervention) and Outcome at 2 months (within 2 weeks post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness | Brain Health
Number analyzed (Participants) | 24 | 28
units on a scale | 5.09 (2.54) | 5.38 (1.62)

ADVERSE EVENTS:
Time Frame: approx 3 months (baseline testing, intervention, plus post-testing)
Arm/Group | Mindfulness | Brain Health
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT02816723/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT02816723/SAP_001.pdf